CLINICAL TRIAL: NCT05177016
Title: Evaluation of Outpatient Hemorrhoidectomies at the Paris Saint Joseph Hospital Group
Acronym: EVHA
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: EVHA
Record Dates: First submitted 2021-12-31; First posted 2022-01-04 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Tripedicular Hemorrhoidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemorrhoidal disease is a frequent and disabling condition that is treated medically and surgically. Tri-pedicular hemorrhoidectomy is the most commonly used surgical technique in France. Due to the restrictive postoperative course (pain, secondary risk of bleeding, asthenia, local care several times a day, transit disorders, urinary disorders, nausea/vomiting), conventional hospitalization was preferred to outpatient surgery until 2015 in our department. The motivation to practice ambulatory surgery is in order to satisfy the patients on the one hand and to improve the economic cost of the management on the other hand. According to the HAS, this is a national priority in order to optimize the supply of care. However, situations such as the absence of an accompanying person, the presence of significant co-morbidities or the use of treatment modifying haemostasis do not allow such surgery to be performed on an outpatient basis. Thanks to the implementation of a dedicated care pathway, outpatient tri-pedicular hemorrhoidectomy at the Paris Saint-Joseph Hospital Group has increased from less than 5% in 2015 to more than 80% in 2021. Outpatient care remains a key criterion for the patient in the context of surgical management.

The objective of this work is to evaluate patient satisfaction with this type of care pathway and to identify the factors associated with dissatisfaction with outpatient care. The secondary objectives are to determine the associated factors of non-satisfaction, the profile of patients for whom outpatient care would not be desirable, to determine the actions to be taken to ensure that outpatient care is provided in the best possible way, to homogenize outpatient care within the department (oral information and written support before the operation, anticipation of postoperative measures (prescriptions and postoperative appointments given during the pre-operative consultation), postoperative liaison file given to the patient on discharge).

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient with an indication for tri-pedicular hemorrhoidectomy
* Patient operated on between January 1, 2020 and December 31, 2020
* French-speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient who objects to the use of his or her data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an indication for tri-pedicular hemorrhoidectomy, operated on between January 1, 2020 and December 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with their outpatient care | Day 1
  This outcome corresponds to the satisfaction rate of patient.

SECONDARY OUTCOMES:
Associated factors of non-satisfaction | Day 1
  This outcome corresponds to the comparison of Satisfaction null or mediocre to good or excellent, No to Yes if it was to be done again in Ambulatory, No to Yes if it was to be advised a hemorrhoidectomy in ambulatory to a relative.
Profile of patients for whom outpatient management would not be desirable | Day 1
  This outcome corresponds to the conversion rate for conventional hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent De Parades, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Vinson Bonnet B, Juguet F; French National Coloproctology Society. Ambulatory proctologic surgery: Recommendations of the French National Coloproctology Society (SNFCP). J Visc Surg. 2015 Dec;152(6):369-72. doi: 10.1016/j.jviscsurg.2015.10.001. Epub 2015 Nov 5. No abstract available. PMID 26547481
- [Background] Soudan D, Fathallah N, de Parades V. [Open haemorrhoidectomy as an ambulatory procedure, is it reasonable?]. Presse Med. 2017 Nov;46(11):1106-1107. doi: 10.1016/j.lpm.2017.08.003. Epub 2017 Sep 14. No abstract available. French. PMID 28919275
- [Background] Moult HP, Aubert M, De Parades V. Classical treatment of hemorrhoids. J Visc Surg. 2015 Apr;152(2 Suppl):S3-9. doi: 10.1016/j.jviscsurg.2014.09.012. Epub 2014 Oct 11. PMID 25311960
- [Background] Vinson-Bonnet B, Higuero T, Faucheron JL, Senejoux A, Pigot F, Siproudhis L. Ambulatory haemorrhoidal surgery: systematic literature review and qualitative analysis. Int J Colorectal Dis. 2015 Apr;30(4):437-45. doi: 10.1007/s00384-014-2073-x. Epub 2014 Nov 28. PMID 25427629